CLINICAL TRIAL: NCT04420702
Title: Diffusion Basis Spectrum Imaging of the Prostate: A Virtual Biopsy to Accurately Diagnose Prostate Cancer
Brief Title: Diffusion Basis Spectrum Imaging of the Prostate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Cancer Society, Inc. (Other); The Foundation for Barnes-Jewish Hospital (Other); Midwest Stone Institute. (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201908215; R01CA258690 (NIH)
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Masking Description: -Dr. Kim will be blinded to the DBSI results at the time of biopsy, but will have the conventional MRI interpretation available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Early Detection Cohort (MRI with DBSI) (Experimental): * Magnetic resonance imaging (MRI) with DBSI analysis prior to prostate biopsy
  * Standard of care prostate biopsy will be performed within 12 weeks of MRI
  * Some participants may go on to receive standard of care radical prostatectomy and those participants may have their prostatectomy specimens scanned via MRI with DBSI imaging
  Interventions: Device: MRI with DBSI analysis
- Active Surveillance Cohort (MRI with DBSI) (Experimental): * Magnetic resonance imaging (MRI) with DBSI analysis prior to prostate biopsy
  * Standard of care prostate biopsy will be performed within 12 weeks of MRI
  * Some participants may go on to receive standard of care radical prostatectomy and those participants may have their prostatectomy specimens scanned via MRI with DBSI imaging
  Interventions: Device: MRI with DBSI analysis

INTERVENTIONS:
Device: MRI with DBSI analysis — -The procedure will take approximately 1 hour of the participant's time

SUMMARY:
Diffusion Basis Spectrum Imaging (DBSI) represents a potential leap forward in improving prostate cancer early detection: a non-invasive and accurate imaging test for clinically significant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age and willing and able to provide informed consent.
* Patients with no prior diagnosis of prostate cancer, who are planning to undergo prostate biopsy as clinical standard of care ("early detection cohort")
* Including those men with:

  * an elevated PSA and no prior biopsy
  * an elevated PSA and a negative prior biopsy
* Patients with a prior diagnosis of prostate cancer, who are currently managed with active surveillance, who are planning to undergo biopsy as clinical standard of care ("active surveillance cohort")

Exclusion Criteria:

* Patients with any clinical contraindication to MRI

  *Including but not limited to:
  * Those with metallic implants, such as pacemakers or implantable cardioverter-defibrillators
  * Those with cochlear implants
  * Those with claustrophobia not relieved with medications (patients with claustrophobia who do not need medications for the scan or whose claustrophobia can be managed with medication, are eligible to participate)
  * Those who cannot lie flat for over 1 hour
* Patients with prior prostate surgery for prostate cancer (e.g. radical prostatectomy, focal ablation)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) comparison from biopsy and DBSI | Up to 12 weeks
  * As a per patient analysis, the investigators will use the highest Gleason score from the biopsy as the reference standard
  * In the per patient analysis, Gleason 7 or greater, will be the cut-off as this will be considered "clinically significant". The investigators will also perform similar analyses with cut-offs of Gleason 4+3=7 or greater, as well as Gleason 6 or greater. This will serve as the sensitivity analysis.
Receiver operating characteristic (ROC) comparison from biopsy to DBSI | Up to 12 weeks
  * As a per patient analysis, the investigators will use the highest Gleason score from the biopsy as the reference standard
  * In the per patient analysis, Gleason 7 or greater, will be the cut-off as this will be considered "clinically significant". The investigators will also perform similar analyses with cut-offs of Gleason 4+3=7 or greater, as well as Gleason 6 or greater. This will serve as the sensitivity analysis.
Prostate sector analysis as measured by comparison of the highest Gleason score from each of the 10 biopsy sectors to the DBSI predicted pathology from each sector | Up to 12 weeks

SECONDARY OUTCOMES:
Comparison of Gleason score from the MRI regions of interest to the DBSI predicted pathology | Up to 12 weeks
  -Only for those patients with a suspicious MRI lesion
Area under the curve (AUC) comparison from DBSI to conventional MRI interpretation | Up to 12 weeks
Receiver operating characteristic (ROC) comparison from DBSI to conventional MRI interpretation | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ippolito, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu